CLINICAL TRIAL: NCT06476847
Title: The Role of Cognitive Biases in the Decision to Request, Offer, Accept and Continue on PrEP From a Health Care Provider and Patient Perspective (Men Who Have Sex With Men)
Brief Title: A Simple Intervention to Increase Persistence on PrEP in MSM to Improve Decision Making
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H-45113; 1K01MH119923-01A1 (NIH)
Record Dates: First submitted 2024-06-21; First posted 2024-06-26 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: HIV Infections
Keywords: Pre-exposure prophylaxis (PrEP); Persistence; Vulnerable populations; Men having sex with men (MSM); South Africa
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants randomized into this group will receive a behavioral economics informed intervention to improve persistence among amongst high risk men newly initiating PrEP in South Africa.
  Interventions: Behavioral: PrEP persistence
- Control group (No Intervention): Usual care for high risk men newly initiating PrEP in South Africa.

INTERVENTIONS:
Behavioral: PrEP persistence — A light touch, once off, low cost. lay counsellor led intervention, designed to focus decision making around HIV prevention addressing present bias, salience and over optimism. The intervention package consists of evidence informed reminders, commitment pledges and planning prompts.
  Arms: Intervention group

SUMMARY:
Oral HIV pre-exposure prophylaxis (PrEP) is a highly effective HIV prevention modality that requires individuals to take a daily tablet to prevent themselves acquiring HIV. In South Africa while this is freely available in the public sector, persistence (that is continuation after initiation) is low amongst vulnerable populations, including men who have sex with men (MSM).

This study is a feasibility and acceptability study of a behavioral economics informed intervention to improve persistence amongst MSM newly initiating PrEP in South Africa. The goal of this study is to show that this approach is possible in a routine setting and gather the necessary data for a fully powered effectiveness trial.

Study participants will complete a baseline questionnaire and then be randomized to either receive standard of care (control) or to receive the intervention. The intervention package consists of evidence informed reminders, commitment pledges and planning prompts. The intervention package aims to address present bias, optimism bias and salience. The intervention is delivered and the enrollment visit and then through mobile phone reminders / text messages. There is no further in person interaction after the initial interaction. Participants may be contacted for a telephonic enplane questionnaire. Outcome data is obtained from passive followup through routine medical record review with the primary end point being persistence at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Not currently on pre exposure prophylaxis (PrEP); no PrEP within the last 12 months
* Initiating PrEP on the date of enrolment
* Access to a mobile phone
* Willing and able to provide written informed consent in English

Exclusion Criteria:

* PrEP status unknown
* Previous PrEP experience within the last year (12 months from enrolment)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2025-01-23 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Target population recruitment (feasibility) | 18 months
  The percent of participants enrolled from those that meet eligibility criteria and are offered will be assessed from screening log.
Fidelity to intervention (feasibility) | 18 months
  Percent of intervention interactions that are delivered in the first 3 months (Max interactions in 3 months = 2 visit reminders and 24 text messages (2 per week) = 26 total interactions).
Acceptability by intervention participants | 18 months
  The percent of participants that accept to participate in the intervention (set reminders/receive text messages) after being randomized to the intervention arm.

SECONDARY OUTCOMES:
PrEP persistence at 3 months, 6 months, and 12 months | 4 months, 7 months, 13 months
  PrEP persistence is defined as having at least a specific number of months of PrEP dispensed after study enrolment. The outcome is determined at the subsequent month to allow for variable timing around return visits.
  For example persistence at 3 months is defined as having at least 90 days of PrEP dispensed by 4 months. Similarly, persistence at 6 months requires 180 days of PrEP dispensed by 7 months and persistence at 12 months requires 360 days of PrEP dispensed by 13 months.

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence C Long, PhD MCom, Principal Investigator — Boston University School of Public Health,Global Health
Locations (2):
- Boston Univeristy School ofPublic Health, Global Health, Boston, Massachusetts, United States
- The Aurum POP INN Clinic, Pretoria, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: No